CLINICAL TRIAL: NCT02036307
Title: Supplementation With Omega-3: Mechanism of Action
Acronym: SOMA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was suspended because there is no more funds to complete the study.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Dhananjay Vaidya, Associate Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NA_00076636
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Hypertriglyceridemia
Keywords: Fish oils; Triglycerides; Blood pressure
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DHA-enriched (Experimental): DHA-enriched supplement (DHA 3g + 600 mg EPA in 6 g of fish oil/day)
  Interventions: Dietary Supplement: DHA-enriched
- EPA-enriched (Experimental): EPA-enriched supplement (EPA 2.4 g + DHA 600mg in 6 g of fish oil/day)
  Interventions: Dietary Supplement: EPA-enriched

INTERVENTIONS:
Dietary Supplement: DHA-enriched — DHA 3g + 600 mg EPA in 6 g of fish oil/day given for 4 weeks
  Other Names: Carlson Labs - Super DHA Gems
  Arms: DHA-enriched
Dietary Supplement: EPA-enriched — EPA 2.4 g + DHA 600mg in 6 g of fish oil/day for 4 weeks
  Other Names: Carlson Labs EPA gems
  Arms: EPA-enriched

SUMMARY:
This is a trial of two marketed fish oil supplements, one with a high EPA:DHA ratio and the other with a high DHA:EPA ratio, to examine differential effects on platelet function, blood pressure, and fasting triglyceride levels.

DETAILED DESCRIPTION:
Observational studies have shown that fish consumption is associated with a lower risk of cardiovascular disease, and clinical trials have demonstrated that fish oil nutritional supplementation is associated with improvement in cardiometabolic risk factor profiles including fasting triglycerides and blood pressure. However, the mechanisms of action of fish oils are not well understood. Specifically, the effects of different compositions in terms of the ratio of the fatty acids EPA and DHA are not known. We are proposing a pilot and feasibility study of fish oil nutritional supplementation in 40 healthy adult participants with two different commercially available fish oil (high EPA/DHA ratio, high DHA/EPA ratio, sample of 20 per group) with the hypothesis that 4 weeks of supplementation with fish oil results in differential changes in platelet function, blood pressure and fasting triglyceride levels . We will also bank blood and urine for future mechanistic studies. This pilot study will allow us to collect preliminary data for definitive mechanistic studies of the effects of fish oil supplementation and to demonstrate the feasibility of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 20-75 years of age.
* Participant of the Principal Investigator's prior studies studies who have agreed to be contacted for future studies.

Exclusion Criteria:

* Current user of fish oil supplements
* Current user of statins
* Allergy to fish or seafood products
* Diagnosed/treated diabetes mellitus
* Using aspirin or NSAIDS or other "blood-thinning medication"

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Fasting triglyceride level | 4 weeks
  Fasting serum triglyceride levels

SECONDARY OUTCOMES:
Seated blood pressure | 4 weeks
  Seated blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Dhananjay Vaidya, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share the individual patient data.